CLINICAL TRIAL: NCT01049347
Title: Hypothalamus-pituitary-adrenal System: Role of the Mineralocorticoid Receptor and Longitudinal Study in Depressed Patients
Brief Title: Amitriptyline and Paroxetine Treatment of Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Prof. Dr. Michael Deuschle, Central Institute of Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AmiPar; DFG De 660/1-1 (Other Grant/Funding Number: German Research Council)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Unipolar Depression
Keywords: depression
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Amitriptyline; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amitriptyline (Active Comparator)
  Interventions: Drug: amitriptyline
- paroxetine (Active Comparator)
  Interventions: Drug: paroxetine

INTERVENTIONS:
Drug: amitriptyline — 150 mg oral, daily, single evening dose, 35 days
  Arms: amitriptyline
Drug: paroxetine — 40 mg oral, single dose, morning, 35 days
  Arms: paroxetine

SUMMARY:
Activation of the hypothalamus-pituitary-adrenal system is monitored using saliva cortisol sampling during the antidepressant treatment with amitriptyline and paroxetine in moderately to severely depressed patients. Additionally, serum and plasma are sampled during the 5-week study period in order to study endocrine and metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* age: above 18
* depression according DSM-IV

Exclusion Criteria:

* bipolar disorder
* substance dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 1997-10; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (21-item version) | baseline, weekly assessments for 5 weeks

SECONDARY OUTCOMES:
cortisol in saliva (8.00, 16.00, 22.00) during wash-out (6 days) and 35 days of treatment | daily during wash-out (days -6 to -1) and active treatment (days 1 to 35)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Deuschle, MD, Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany

REFERENCES:
- [Derived] Schilling C, Gilles M, Blum WF, Daseking E, Colla M, Weber-Hamann B, Lederbogen F, Krumm B, Heuser I, Wudy SA, Kopf D, Deuschle M. Leptin plasma concentrations increase during antidepressant treatment with amitriptyline and mirtazapine, but not paroxetine and venlafaxine: leptin resistance mediated by antihistaminergic activity? J Clin Psychopharmacol. 2013 Feb;33(1):99-103. doi: 10.1097/JCP.0b013e31827cb179. PMID 23277262
- [Derived] Paslakis G, Kopf D, Westphal S, Gilles M, Lederbogen F, Hamann B, Heuser I, Deuschle M. Treatment with paroxetine, but not amitriptyline, lowers levels of lipoprotein(a) in patients with major depression. J Psychopharmacol. 2011 Oct;25(10):1344-6. doi: 10.1177/0269881110382469. Epub 2010 Oct 15. PMID 20952454